CLINICAL TRIAL: NCT06379399
Title: Trifluridine/Tipiracil Combined With Cetuximab in the Treatment of Third-line and Above RAS/BRAF Wild-type Metastatic Colorectal Cancer: A Single-center, Prospective Phase Ib/II Study
Brief Title: Trifluridine/Tipiracil Combined With Cetuximab in the Treatment of Third-line and Above RAS/BRAF Wild-type mCRC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wangxia LV (Other)
Responsible Party: Sponsor-Investigator, Wangxia LV, Deputy Director of Colorectal Medicine, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-1072
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer Metastatic
Keywords: RAS/BRAF wild-type
MeSH Terms: interventions — Cetuximab; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cetuximab Combined With Trifluridine/Tipiracil (Experimental)
  Interventions: Drug: Cetuximab; Drug: Trifluridine/Tipiracil

INTERVENTIONS:
Drug: Cetuximab — Cetuximab will be administered at a fixed dose of 500 mg/m2 once every 2 weeks;
  Other Names: Erbitux
Drug: Trifluridine/Tipiracil — Phase I:
  1. 6 patients (male and female) will be enrolled to evaluate safety. Patients will receive Trifluridine/Tipiracil at a dose of 35mg/m2 (maximum single dose of 80 mg). Patients will be followed up for Dose-Limiting Toxicities (DLTs) (2 Cycles, Day 1-Day 28). If ≤2 patients experience DLTs (2 Cycles, Day 1-Day 28), the study will proceed to Phase II with a dose of 35mg/m2. If ≥3 patients experience DLTs (2 Cycles, Day 1-Day 28), the study will proceed to Phase II with a dose of 30mg/m2.
  2. Based on the results of the 35mg/m2 dose group, 6 patients (male and female) will be enrolled in the 30mg/m2 dose group to evaluate safety. Patients will be followed up for DLTs (2 Cycles, Day 1-Day 28). If ≤2 patients experience DLTs (1 Cycle, Day 1-Day 28), the study will proceed with a dose of 30mg/m2 in Phase II.
  Phase II:
  Trifluridine/Tipiracil: po, twice daily from Day 1-5, every two weeks, based on the recommended dose from Phase I;
  Other Names: TAS-102; FTP/TPI

SUMMARY:
This study is a single-center, prospective, single-arm exploratory study aimed at evaluating the efficacy and safety of trifluridine/tipiracil in combination with cetuximab in the treatment of third-line and above RAS/BRAF wild-type metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient able and willing to provide written informed consent and to comply with the study protocol and follow-up inspection.
2. Histologically or cytologically confirmed metastatic adenocarcinoma of the colon; excluding appendiceal and anal canal cancers.
3. Previously received at least second-line treatment, including two standard treatment regimens (such as fluoropyrimidine, capecitabine, irinotecan, oxaliplatin with or without anti-VEGF or anti-EGFR agents), if previously received first-line anti-EGFR therapy, achieving at least a partial response (PR) or above, with a discontinuation interval of at least one year.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) (based on RECIST 1.1 criteria, with the longest diameter of tumor lesions on CT/MRI scan ≥10mm, and the shortest diameter of lymph node lesions on CT/MRI scan ≥15mm).
6. Wild-type RAS/BRAF gene detected.
7. Able to take oral medication.
8. Normal organ function, meeting the following criteria within 14 days before treatment initiation:

   * Neutrophil count ≥1.5×10^9/L;
   * Platelet count ≥75×10^9/L;
   * Hemoglobin ≥9.0g/dL;
   * Aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN) (or ≤5×ULN if liver metastases);
   * Alanine aminotransferase (ALT) ≤2.5×ULN (or ≤5×ULN if liver metastases);
   * Total bilirubin ≤1.5×ULN;
   * Creatinine clearance (calculated by Cockcroft and Gault formula) >60mL/min or serum creatinine ≤1.5×ULN;
9. Expected survival time >3 months (90 days).
10. Women of childbearing potential must have used reliable contraception for 7 days prior to enrollment, have had a negative pregnancy test, and agree to use appropriate contraception methods during the trial and for 6 months after the last dose of investigational drug. Men must agree to use appropriate contraception methods or have undergone surgical sterilization during the trial and for 6 months after the last dose of investigational drug.

Exclusion Criteria:

1. Prior treatment with Trifluridine/Tipiracil;
2. Patients with known dMMR or MSI-H advanced colorectal cancer who have not previously received anti-PD-1 or PD-L1 inhibitors;
3. Participation in another drug clinical trial or receipt of systemic chemotherapy, radiotherapy, or biologic therapy within the past 4 weeks;
4. Known or suspected brain metastases;
5. Synchronous or metachronous cancer with a disease-free survival of ≥5 years (except for colorectal cancer) excluding cured or curatively treated mucosal cancers (esophageal cancer, gastric cancer, cervical cancer, non-melanoma skin cancer, bladder cancer, etc.);
6. Factors significantly affecting oral drug absorption, such as dysphagia, chronic diarrhea, and gastrointestinal obstruction; uncontrolled Crohn's disease or ulcerative colitis;
7. Symptomatic malignant effusion requiring symptomatic treatment (including pleural effusion, ascites, pericardial effusion);
8. Pregnant or lactating women; patients with reproductive potential unwilling or unable to use effective contraceptive measures;
9. Known allergy to the investigational drug, drug class, or its components;
10. Requirement for systemic corticosteroid therapy (excluding local steroids and cetuximab pre-treatment);
11. History of interstitial lung disease (interstitial pneumonia, pulmonary fibrosis, etc.) or radiographic evidence of interstitial lung disease;
12. Active local or systemic infections requiring treatment;
13. New York Heart Association (NYHA) functional classification ≥II or severe heart disease;
14. Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) or history of active hepatitis B or hepatitis C;
15. Unresolved toxicity (CTCAE>Grade 1) or incomplete recovery from previous cancer surgery.
16. Patients deemed unsuitable for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 12 months
  Progression-free survival defined as the time elapsed between the randomization and the date of radiologic tumour progression according to RECIST version 1.1 by investigator's judgement or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 12 months
  Overall survival defined as the observed time elapsed between the date of first treatment and the date of death due to any cause.
Overall Response Rate (ORR) | Approximately 12 months
  Objective Response Rate defined as the proportion of patients with objective evidence of complete response (CR) or partial response (PR) according to RECIST version 1.1 criteria and using investigator's tumor assessment.
Disease Control Rate( DCR) | Approximately 12 months
  Disease Control Rate defined as the proportion of patients with objective evidence of CR or PR or stable disease (SD) according to RECIST version 1.1 criteria and using investigator's tumor assessment.
Quality of life: EORTC QLQ-C30 | Approximately 12 months
  Assess patients health and activities using the European Organization for Research and Treatment of Cancer Core Quality of Life (EORTC QLQ-C30) module.
Adverse Events(safety) | Up to 28 days after discontinuation of study drug or start of subsequent therapy.
  Adverse events were recorded according to Common Terminology Criteria for Adverse Events (version 5.0) of the National Cancer Institute that participants received at least one dose of protocol treatment after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Lv, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No